CLINICAL TRIAL: NCT01141855
Title: Effectiveness of Inpatient Initiated Varenicline Tartrate for Smoking Cessation, for Smoking Related Illnesses.
Brief Title: Smoking Termination Opportunity for inPatients
Acronym: STOP
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The Queen Elizabeth Hospital (Other)
Responsible Party: Associate Professor Brian James Smith, The Queen Elizabeth Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 2008012
Record Dates: First submitted 2010-06-10; First posted 2010-06-11 (Estimated); Last update posted 2012-08-08 (Estimated); Status verified 2010-04

CONDITIONS: Tobacco Use Disorder
Keywords: Cardiovascular Diseases; Peripheral Vascular Diseases; Cerebrovascular Stroke; Lung Diseases, Obstructive; Asthma; Tobacco Use Disorder; Smoking; Smoking Cessation
MeSH Terms: conditions — Tobacco Use Disorder; Cardiovascular Diseases; Peripheral Vascular Diseases; Stroke; Lung Diseases, Obstructive; Asthma; Smoking; Smoking Cessation | interventions — Varenicline; Counseling

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Champix plus counselling (Experimental): varenicline tartrate will be initiated whilst subjects are inpatients with the standard MIMS dosing schedule (including period of titration). In combination with Quit SA (5A) telephone counselling service
  Interventions: Drug: Champix
- counselling alone (Active Comparator): 5A counselling via Quit SA (quitline) telephone counselling service. (maximum 8 phone calls per subject within a 3 month period).
  Interventions: Behavioral: Counselling alone

INTERVENTIONS:
Drug: Champix — Standard MIMS dosage (including period of titration) will be used. 0.5mg daily for 3 days 0.5mg b.d. for 4 days
  1mb b.d. for 70 days (full course 3 months)
  Other Names: varenicline tartrate; Chantix
  Arms: Champix plus counselling
Behavioral: Counselling alone — Quit SA 5A counselling over the phone. Maximum 8 calls over a 3 month period
  Other Names: Quitline counselling service
  Arms: counselling alone

SUMMARY:
The Smoking Termination Opportunity for inPatients, (STOP) project is designed to capture the opportunity that is provided by admission for acute smoking related illness, to assist patients through withdrawal by use of a combination of:

* the new medication Champix with
* best practice counselling
* initiated in an inpatient setting

to achieve:

* sustained smoking abstinence
* reduced hospital bed and health service utilisation
* reduced inpatient smoking and craving prior to discharge

DETAILED DESCRIPTION:
A national standard in public hospitals for the management of smoking in patients admitted with smoking related acute illnesses is lacking. Where such patients have continued to smoke up until the time of admission, it can be assumed that "primary" prevention has failed.

Once admitted, there is a vastly under-utilised opportunity, by use of a structured and systematic approach, to intervene with a secondary prevention attempt. This takes advantage of the synergy of:

1. the smoker is a "captive audience" and may be receptive to considering lifestyle factors that have lead to the admission, and
2. best practice medication and counselling can be initiated prior to discharge. If proven to be cost-effective in our analysis, a systematic roll-out of this secondary prevention initiative would be advocated. ie translation of research into practice.

ELIGIBILITY:
Inclusion Criteria:

* Smoker of at least 10 cigarettes per day on average over the past 12 months
* Inpatient with an anticipation admission of at least one day
* Willingness to quit smoking
* Aged between 20 and 75 years
* A plan of discharge to go home
* Acute hospital admission with cardiovascular, cerebrovascular, peripheral vascular diseases or airways (asthma and/or Chronic Obstructive Pulmonary disease

Exclusion Criteria:

* Subject preference to use an alternative pharmacotherapy for smoking cessation
* Respiratory patient being considered for home oxygen
* Pregnancy
* Breast feeding
* Acute or pre-existing severe psychiatric illnesses
* Past history of psychosis or suicidal ideation
* Renal impairment with creatinine clearance <30ml/min

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Actual)
Dates: Start 2008-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Smoking abstinence | one year
  Continued smoking abstinence is defined as: less than or equal to no more than 5 cigarettes smoked during the period of 2 weeks to 12 months post enrollment.

SECONDARY OUTCOMES:
Reduced hospital bed utilisation | one year
  Hospital casemix/DRG data will be collected for the 5 years prior to enrollment and one year post enrollment. This will be supplemented by SA Department of Health data and PBS/MBS data sets of study completion, to monitor admissions at other hospitals and GP visits.
7-day point prevalence | from 2 weeks to 3 months post enrollment
  Defined as no cigarettes for the previous 7 days
Reduction in health care costs | one year
  Reduced health care costs with greater economic value will be relative to other health interventions. Four seperate economic models will be built for vascular diseases: cardiovascular, cerebrovascular and peripheral vascular diseases and airways diseases: asthma and/or chronic obstructive pulmonary disease. Each model will compare outcomes and costs for varenicline and counselling compared to counselling alone, and will incorporate epidemiological data on natural disease progression of smokers and previous smokers from the four disease profiles split by gender if indicated.
Inpatient craving levels | baseline to end of inpatient stay
  Craving scales will be used to assess levels during inpatient stay (pre and post intervention delivery)
Prevalence of inpatient smoking | From baseline to end of inpatient stay
  Measured by self-report and observation by hospital and study staff prior to discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Brian J Smith, MBBS; FRACP;PhD;Dip Clin Epid, Principal Investigator — The Queen Elizabeth Hospital
Locations (3):
- Australia (3):
  - Royal Adelaide Hospital, Adelaide, South Australia
  - The Queen Elizabeth Hospital, Adelaide, South Australia
  - Lyell McEwin Health Service, Adelaide, South Australia

REFERENCES:
- [Derived] Smith BJ, Carson KV, Brinn MP, Labiszewski NA, Peters MJ, Fitridge R, Koblar SA, Jannes J, Veale AJ, Goldsworthy SJ, Litt J, Edwards D, Esterman AJ. Smoking Termination Opportunity for inPatients (STOP): superiority of a course of varenicline tartrate plus counselling over counselling alone for smoking cessation: a 12-month randomised controlled trial for inpatients. Thorax. 2013 May;68(5):485-6. doi: 10.1136/thoraxjnl-2012-202484. Epub 2012 Sep 19. PMID 22993168